CLINICAL TRIAL: NCT07177391
Title: Discontinuous Echocardiographic Subcostal Cardiac Output Measurement by the Right Ventricular Outflow Tract in Critical Care
Brief Title: Discontinuous Echocardiographic Subcostal Cardiac Output Measurement
Acronym: RIGHT WAY
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2024/0200/OB; 2024-A01706-41 (Other: ANSM)
Record Dates: First submitted 2025-09-09; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Cardiac Output Measurement
Keywords: diagnosis of circulatory failure; multiple failures in critical care

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Discontinuous subcostal echocardiographic cardiac output assessment — Right Ventricular Outflow Chamber Diameter (RVOD) and Left Ventricular Outflow Chamber Diameter (LVOD) assessments via subcostal approach

SUMMARY:
Cardiac output (CO) monitoring is recommended for the most serious and multiple-failure patients in critical care and allows the diagnosis of acute circulatory failure as well as its etiology and also allows the monitoring of treatments. However, although allowing an adaptation of hemodynamic treatments and being integrated into a therapeutic personalization approach in situations of acute circulatory failure, the measurement of CO is conditioned by the availability of devices, by their sometimes problematic invasiveness, as well as their cost. In addition, the discontinuous measurement of CO by echocardiography is made difficult in the context of resuscitation with patients who are less mobilizable and less echogenic.

DETAILED DESCRIPTION:
The subcostal assessment route is the classic emergency route. It allows for the analysis of the basic segmental kinetics of the left ventricle, an analysis of the Left Ventricular Ejection Fraction (LVEF), the search for pericardial effusion or even tamponade, or the search for right ventricular dilation. A measurement of CO via the right ventricular outflow tract using transthoracic echocardiography has never been described in the literature, although it is feasible, based on the same mathematical rationale as the standard measurement of cardiac output via the left ventricular outflow tract (which takes into account the diameter of the outflow tract and the subvalvular time-velocity integral [TVI]).

Since at all times the left (systemic) CO is equal to the right (venous return) CO, it is therefore possible to consider a measurement of CO via the subcostal route. By not complicating the standard care of patients in critical care, especially in situations of acute circulatory failure, and by adding only a few seconds or even minutes to an examination already recommended and routine in critical care, this evaluation approach seems interesting given the need and the recommendations in force on the monitoring of patients in intensive care and more particularly of DC.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (Age ≥ 18 years)
* Patient admitted to the intensive care unit at Rouen University Hospital.
* Transthoracic echocardiography (TTE) is required upon admission or during the patient's stay for diagnostic assessment and/or therapeutic monitoring.

Exclusion Criteria:

* Person deprived of liberty by an administrative or judicial decision or person placed under judicial protection/guardianship or curatorship
* Patient not affiliated with the social security system
* Refusal by the patient or trusted person if the patient is incapable of expressing consent
* Pregnant woman
* Dying patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective cohort including patients admitted to the intensive care unit of the Rouen University Hospital and requiring, upon admission or during their stay, the performance of a transthoracic echocardiography for diagnostic assessment and/or therapeutic monitoring.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2025-09-09 (Actual); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Measurement of Cardiac Output (CO) via the subcostal route | At Enrollment visit and DAY 28
  To assess the concordance of the measurement of cardiac output in the ejection chamber of the right ventricle (DC-CEVD, innovative method) with that of cardiac output in the ejection chamber of the left ventricle (DC-CEVG, reference method) on subcostal transthoracic ultrasound (TTE).

SECONDARY OUTCOMES:
Compare the measurement success rate of DC-CEVD to that of DC-CEVG. | At Enrollment visit and DAY 28
  Evaluate the success of cardiac output measurement, defined by the fact of rendering a flow measurement
To assess the concordance of DC variation during preload-dependence search maneuvers (passive leg raise) in intubated and ventilated patients between DC-CEVD and DC-CEVG measurements. | At Enrollment visit and DAY 28
  Evaluation of DC Variation during the preload-dependence search maneuver: passive leg raise test and 1-minute DC measurement according to the two modalities (DC-CEVD and DC-CEVG measurements).
DC measurement by transpulmonary thermodilution device | At Enrollment visit and DAY 28
  Search for the best concordance of the DC-CEVD to the Plan for Continuity of Circulation and Oxygenation (PCCO) and of the DC-CEVG to the PCCOi in a patient who has a transpulmonary thermodilution device with analysis of the pulse wave contour (PCCO), (PiCCO2),

CONTACTS AND LOCATIONS:
Locations (1):
- University Rouen Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No
The data provided will be the property of the sponsor and will be used solely for its own research activities.